CLINICAL TRIAL: NCT00483938
Title: The Individualized Management With Pegasys and Ribavirin Offering Viral Eradication (IMPROVE) Trial
Brief Title: The Individualized Management With Pegylated-interferon Alfa-2a (Pegasys) and Ribavirin (Copegus) Offering Viral Eradication: A Study of Pegylated-interferon Alfa-2a Plus Ribavirin in Participants With Chronic Hepatitis C (CHC) Non-genotype 2/3 (IMPROVE)
Acronym: IMPROVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21035
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (7):
- Pegylated-interferon Alfa-2a + Ribavirin (Group A) (Experimental): Participants with HCV RNA levels greater than (>) 15 international units per milliliter (IU/mL) at Week 4, HCV RNA greater than or equal to (>=) 15 IU/mL at Week 8, and either HCV RNA less than (<) 15 IU/mL or >=2 times logarithmic (2 log10) drop at Week 12, will receive pegylated-interferon alfa-2a (Pegasys) 180 micrograms (mcg) subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 milligrams (mg) orally daily for 48 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin
- Pegylated-interferon Alfa-2a + Ribavirin (Group B) (Experimental): Participants with HCV RNA levels >15 IU/mL at Week 4, HCV RNA >=15 IU/mL at Week 8, and either HCV RNA <15 IU/mL or >=2 log10 drop at Week 12, will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 72 weeks, and ribavirin 1000 to 1400 mg orally daily for 72 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin
- Pegylated-interferon Alfa-2a + Ribavirin (Group C) (Experimental): Participants with HCV-RNA levels >15 IU/mL at Week 4, and HCV-RNA <15 IU/mL at Week 8, will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 36 weeks, and ribavirin 1000 to 1400 mg orally daily for 36 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin
- Pegylated-interferon Alfa-2a + Ribavirin (Group D) (Experimental): Participants with HCV-RNA levels >15 IU/mL at Week 4, and HCV-RNA <15 IU/mL at Week 8, will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 mg orally daily for 48 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin
- Pegylated-interferon Alfa-2a + Ribavirin (Group E) (Experimental): Participants with HCV-RNA levels <15 IU/mL at Week 4, will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 24 weeks, and ribavirin 1000 to 1400 mg orally daily for 24 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin
- Pegylated-interferon Alfa-2a + Ribavirin (Group F) (Experimental): Participants with HCV-RNA levels <15 IU/mL at Week 4, will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 mg orally daily for 48 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin
- Pegylated-interferon Alfa-2a + Ribavirin (Group NR) (Experimental): Participants who do not have any change in HCV-RNA levels at Weeks 4, 8, and 12 will not be randomized (NR) to any of the other groups. Participants will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 mg orally daily for 48 weeks.
  Interventions: Drug: Pegylated-interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated-interferon Alfa-2a — Participants will receive pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for the specified duration.
  Other Names: Pegasys
Drug: Ribavirin — Participants will receive ribavirin 1000 to 1400 mg orally daily for the specified duration.
  Other Names: Copegus

SUMMARY:
This study will compare the efficacy and safety of treatment with pegylated-interferon alfa-2a plus ribavirin in participants with non-genotype 2/3 CHC who, after 12 weeks of study treatment, have undetectable hepatitis C virus (HCV)-ribonucleic acid (RNA) or a greater than or equal to (>=) 2 log10 drop in HCV-RNA. Participants will be randomized to receive pegylated-interferon alfa-2a 180 micrograms subcutaneously weekly plus ribavirin (1000-1400 milligram [mg]) orally daily for the specified duration, followed by 24 weeks of treatment-free follow-up. Participants with detectable HCV-RNA and less than (<) 2 log10 drop in HCV-RNA at week 12 will discontinue therapy.

ELIGIBILITY:
Inclusion Criteria:

* evidence of CHC;
* evidence of hepatitis C non-genotype 2 or 3;
* compensated liver disease.

Exclusion Criteria:

* infection with HCV genotype 2 or 3;
* history of having received systemic antiviral therapy with activity against CHC <=3 months prior to start of study;
* hepatitis A, hepatitis B or human immunodeficiency virus (HIV) infection;
* history or evidence of a medical condition associated with chronic liver disease other than CHC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Milwaukee, Wisconsin, United States
- Canada (17):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Vancouver, British Columbia
  - Vernon, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - East York, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Woodbridge, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Lee SS, Sherman M, Ramji A, Greenbloom S, Elkashab M, Pluta H, Hilzenrat N, Balshaw R, Usaty C, Myers RP. Randomised clinical trial: the efficacy of treatment, guided by a shorter duration of response, using peginterferon alfa-2a plus ribavirin for hepatitis C virus other than genotypes 2 or 3. Aliment Pharmacol Ther. 2012 Jan;35(1):37-47. doi: 10.1111/j.1365-2036.2011.04911.x. Epub 2011 Nov 2. PMID 22050141

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegylated-interferon Alfa-2a + Ribavirin (Group A): Participants with hepatitis C virus (HCV) ribonucleic acid (RNA) levels greater than (>) 15 international units per milliliter (IU/mL) at Week 4, HCV RNA greater than or equal to (>=) 15 IU/mL at Week 8, and either HCV RNA less than (<) 15 IU/mL or >=2 times logarithmic (2 log10) drop at Week 12, received pegylated-interferon alfa-2a (Pegasys) 180 micrograms (mcg) subcutaneously once in a week for 48 weeks, and ribavirin (Copegus) 1000 to 1400 milligrams (mg) orally daily for 48 weeks.
- Pegylated-interferon Alfa-2a + Ribavirin (Group B): Participants with HCV RNA levels >15 IU/mL at Week 4, HCV RNA >=15 IU/mL at Week 8, and either HCV RNA <15 IU/mL or >=2 log10 drop at Week 12, received pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 72 weeks, and ribavirin 1000 to 1400 mg orally daily for 72 weeks.
- Pegylated-interferon Alfa-2a + Ribavirin (Group C): Participants with HCV-RNA levels >15 IU/mL at Week 4, and HCV-RNA <15 IU/mL at Week 8, received pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 36 weeks, and ribavirin 1000 to 1400 mg orally daily for 36 weeks.
- Pegylated-interferon Alfa-2a + Ribavirin (Group D): Participants with HCV-RNA levels >15 IU/mL at Week 4, and HCV-RNA <15 IU/mL at Week 8, received pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 mg orally daily for 48 weeks.
- Pegylated-interferon Alfa-2a + Ribavirin (Group E): Participants with HCV-RNA levels <15 IU/mL at Week 4, received pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 24 weeks, and ribavirin 1000 to 1400 mg orally daily for 24 weeks.
- Pegylated-interferon Alfa-2a + Ribavirin (Group F): Participants with HCV-RNA levels <15 IU/mL at Week 4, received pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 mg orally daily for 48 weeks.
- Pegylated-interferon Alfa-2a + Ribavirin (Group NR): Participants who did not have any change in HCV-RNA levels at Weeks 4, 8, and 12 were not randomized (NR) to any of the other groups. Participants received pegylated-interferon alfa-2a 180 mcg subcutaneously once in a week for 48 weeks, and ribavirin 1000 to 1400 mg orally daily for 48 weeks.
Period: Overall Study
Arm/Group | Pegylated-interferon Alfa-2a + Ribavirin (Group A) | Pegylated-interferon Alfa-2a + Ribavirin (Group B) | Pegylated-interferon Alfa-2a + Ribavirin (Group C) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) | Pegylated-interferon Alfa-2a + Ribavirin (Group F) | Pegylated-interferon Alfa-2a + Ribavirin (Group NR)
Started | 41 | 43 | 30 | 31 | 25 | 26 | 40
Completed | 36 | 24 | 30 | 25 | 23 | 18 | 0
Not Completed | 5 | 19 | 0 | 6 | 2 | 8 | 40
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 6 | 0 | 0 | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0 | 2 | 1 | 1 | 3
Not completed — Death | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 9 | 0 | 4 | 0 | 4 | 32

BASELINE CHARACTERISTICS:
Population: The safety (SAF) population included participants who received at least one dose of study medication and had at least one post-baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegylated-interferon Alfa-2a + Ribavirin (Group A) | Pegylated-interferon Alfa-2a + Ribavirin (Group B) | Pegylated-interferon Alfa-2a + Ribavirin (Group C) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) | Pegylated-interferon Alfa-2a + Ribavirin (Group F) | Pegylated-interferon Alfa-2a + Ribavirin (Group NR) | Total
Number analyzed (Participants) | 41 | 43 | 30 | 31 | 25 | 26 | 40 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (8.55) | 51.0 (7.39) | 48.7 (11.54) | 47.8 (9.16) | 47.0 (10.38) | 47.0 (9.76) | 51.7 (7.52) | 49.5 (9.13)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 19 | 10 | 12 | 6 | 9 | 13 | 85
  Male | 25 | 24 | 20 | 19 | 19 | 17 | 27 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response (SVR) (Groups A and B)
Description: SVR was defined as success if the participant had HCV RNA levels <15 IU/mL as measured by COBAS AmpliPrep/COBAS TaqMan® HCV test at the 24-week untreated follow-up visit (HCV-RNA levels obtained at least 18 weeks after last dose of either pegylated-Interferon alfa-2a or ribavirin were considered if the 24-week untreated follow-up visit data were missing). Percentage of participants with SVR for Groups A and B was reported in this analysis.
Time Frame: At 24-week untreated follow-up visit (up to 72 weeks for Group A, up to 96 weeks for Group B)
Population: Intent-to-treat (ITT) population included randomized participants who received at least one dose of study medication and who had a baseline HCV-RNA which was at least 15 IU/mL. Here, "Number of Participants Analyzed" = the participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated-interferon Alfa-2a + Ribavirin (Group A) | Pegylated-interferon Alfa-2a + Ribavirin (Group B)
Number analyzed (Participants) | 41 | 43
percentage of participants | 48.8 | 39.5
Statistical Analysis 1: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group A) vs Pegylated-interferon Alfa-2a + Ribavirin (Group B); SVR: Group A versus Group B; Test type: Superiority or Other; p = 0.510, Fisher Exact

2. Secondary Outcome: Percentage of Participants With SVR (Groups C, D, E, and F)
Description: SVR was defined as success if the participant had HCV RNA levels <15 IU/mL as measured by COBAS AmpliPrep/COBAS TaqMan® HCV test at the 24-week untreated follow-up visit (HCV-RNA levels obtained at least 18 weeks after last dose of either pegylated-Interferon alfa-2a or ribavirin were considered if the 24-week untreated follow-up visit data were missing). Percentage of participants with SVR for Groups C, D, E, and F was reported in this analysis.
Time Frame: At 24-week untreated follow-up visit (up to 60, 72, 48, and 72 weeks for Groups C, D, E, and F, respectively)
Population: ITT. Here, "Number of Participants Analyzed" = the participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated-interferon Alfa-2a + Ribavirin (Group C) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) | Pegylated-interferon Alfa-2a + Ribavirin (Group F)
Number analyzed (Participants) | 30 | 31 | 25 | 25
percentage of participants | 73.3 | 74.2 | 84.0 | 84.0
Statistical Analysis 1: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group C) vs Pegylated-interferon Alfa-2a + Ribavirin (Group D); SVR: Group C versus Group D; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group E) vs Pegylated-interferon Alfa-2a + Ribavirin (Group F); SVR: Group E versus Group F; Test type: Superiority or Other; p = 1.000, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Virological Responses (Groups A, B, C, D, E, and F)
Description: End of treatment response (ETR) was defined as "Success" if the HCV-RNA levels were <15 IU/mL at the end of treatment. Early virological response (EVR) was defined as >=2 log10 decrease in serum HCV RNA or undetectable serum HCV RNA (<15 IU/mL) at Week 12. Complete EVR was defined as "Success", if the HCV-RNA levels were <15 IU/mL at Week 12. Partial EVR was defined as "Success", if there was a >=2 log10 drop in HCV-RNA at Week 12 compared to baseline but with a level that was still >=15 IU/mL at that time point.
Time Frame: Week 12 (Groups C, D, E, and F), and end of treatment (Weeks 48, 72, 36, 48, 24, and 48 for Groups A, B, C, D, E, and F, respectively)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated-interferon Alfa-2a + Ribavirin (Group A) | Pegylated-interferon Alfa-2a + Ribavirin (Group B) | Pegylated-interferon Alfa-2a + Ribavirin (Group C) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) | Pegylated-interferon Alfa-2a + Ribavirin (Group F)
Number analyzed (Participants) | 41 | 43 | 30 | 31 | 25 | 25
percentage of participants
  ETR | 80.5 | 76.7 | 96.7 | 90.3 | 92.0 | 100.0
  Complete EVR | 0 | 0 | 93.3 | 96.8 | 88.0 | 92.0
  Partial EVR | 0 | 0 | 0 | 3.2 | 0 | 0
Statistical Analysis 1: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group A) vs Pegylated-interferon Alfa-2a + Ribavirin (Group B); ETR: Group A versus Group B; Test type: Superiority or Other; p = 0.792, Fisher Exact
Statistical Analysis 2: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group C) vs Pegylated-interferon Alfa-2a + Ribavirin (Group D); ETR: Group C versus Group D; Test type: Superiority or Other; p = 0.612, Fisher Exact
Statistical Analysis 3: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group E) vs Pegylated-interferon Alfa-2a + Ribavirin (Group F); ETR: Group E versus Group F; Test type: Superiority or Other; p = 0.490, Fisher Exact
Statistical Analysis 4: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group C) vs Pegylated-interferon Alfa-2a + Ribavirin (Group D); Complete EVR: Group C versus Group D; Test type: Superiority or Other; p = 0.363, Fisher Exact
Statistical Analysis 5: Comparison: Pegylated-interferon Alfa-2a + Ribavirin (Group E) vs Pegylated-interferon Alfa-2a + Ribavirin (Group F); Complete EVR: Group E versus Group F; Test type: Superiority or Other; p = 1.000, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline up to 96 weeks
Description: Safety population
Arm/Group | Pegylated-interferon Alfa-2a + Ribavirin (Group A) | Pegylated-interferon Alfa-2a + Ribavirin (Group B) | Pegylated-interferon Alfa-2a + Ribavirin (Group C) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) | Pegylated-interferon Alfa-2a + Ribavirin (Group F) | Pegylated-interferon Alfa-2a + Ribavirin (Group NR)
Serious Adverse Events (participants affected / at risk) | 4/41 | 6/43 | 5/30 | 4/31 | 0/25 | 4/26 | 3/40
Other Adverse Events (participants affected / at risk) | 39/41 | 43/43 | 30/30 | 31/31 | 25/25 | 25/26 | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated-interferon Alfa-2a + Ribavirin (Group A) (N=41) | Pegylated-interferon Alfa-2a + Ribavirin (Group B) (N=43) | Pegylated-interferon Alfa-2a + Ribavirin (Group C) (N=30) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) (N=31) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) (N=25) | Pegylated-interferon Alfa-2a + Ribavirin (Group F) (N=26) | Pegylated-interferon Alfa-2a + Ribavirin (Group NR) (N=40)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Emotional/mental (depression, anxiety, irritability, forgetfulness, confusion, anger) (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — This was reported as 'adverse event (AE) cluster' i.e. combination of multiple AEs and not as separate AE preferred terms (PTs).
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 0 | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated-interferon Alfa-2a + Ribavirin (Group A) (N=41) | Pegylated-interferon Alfa-2a + Ribavirin (Group B) (N=43) | Pegylated-interferon Alfa-2a + Ribavirin (Group C) (N=30) | Pegylated-interferon Alfa-2a + Ribavirin (Group D) (N=31) | Pegylated-interferon Alfa-2a + Ribavirin (Group E) (N=25) | Pegylated-interferon Alfa-2a + Ribavirin (Group F) (N=26) | Pegylated-interferon Alfa-2a + Ribavirin (Group NR) (N=40)
Anemia (Blood and lymphatic system disorders) | 12 | 16 | 5 | 7 | 4 | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 9 | 9 | 8 | 3 | 6 | 9 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1 | 1 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 1 | 1 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2 | 2 | 2 | 1 | 0 | 0
Dry eye (Eye disorders) | 3 | 0 | 2 | 2 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 3 | 2
Gastrointestinal symptoms (diarrhea, bloating, gas) (Gastrointestinal disorders) | 14 | 9 | 12 | 11 | 1 | 6 | 4 — This was reported as 'AE cluster' i.e. combination of multiple AEs and not as separate AE PTs.
Nausea (Gastrointestinal disorders) | 11 | 10 | 5 | 8 | 7 | 4 | 5
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 3 | 1 | 2 | 2 | 2
Asthenia (General disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 18 | 22 | 15 | 8 | 10 | 12 | 6
Feeling abnormal (General disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 0
Flu-like symptoms (fever, chills, headache, aches/pains) (General disorders) | 37 | 32 | 23 | 24 | 16 | 21 | 28 — This was reported as 'AE cluster' i.e. combination of multiple AEs and not as separate AE PTs.
Ear infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 3 | 0 | 3 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 4 | 0 | 2 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 2 | 0 | 0 | 1 | 3 | 0
Weight decreased (Investigations) | 3 | 2 | 2 | 3 | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 5 | 4 | 3 | 4 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 1 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2 | 1 | 1 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 7 | 3 | 5 | 1 | 3 | 2
Dysgeusia (Nervous system disorders) | 1 | 2 | 2 | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 5 | 1 | 7 | 0 | 2 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 3 | 3 | 0 | 3
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 0
Emotional/mental (depression, anxiety, irritability, forgetfulness, confusion, anger) (Psychiatric disorders) | 21 | 25 | 15 | 17 | 11 | 15 | 13 — This was reported as 'AE cluster' i.e. combination of multiple AEs and not as separate AE PTs.
Insomnia (Psychiatric disorders) | 16 | 18 | 10 | 6 | 4 | 11 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 7 | 3 | 3 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 6 | 4 | 3 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6 | 0 | 2 | 2 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 9 | 8 | 1 | 4 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 1 | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 1
Skin (injection site reactions, rashes, pruritus) (Skin and subcutaneous tissue disorders) | 24 | 24 | 20 | 16 | 12 | 18 | 16 — This was reported as 'AE cluster' i.e. combination of multiple AEs and not as separate AE PTs.
Hot flush (Vascular disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.